CLINICAL TRIAL: NCT06384105
Title: Prospective Multicentric Study of the Patient Radiation Dose During Five Endourological Procedures: Insertion and Replacement of Ureteral Stent, URS, (Mini-)PCNL/ PCNL and ESWL/SWL
Brief Title: Study of the Patient Radiation Dose During Five Endourological Procedures
Acronym: PRDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Vincent De Coninck, Principal Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRDE1
Record Dates: First submitted 2024-04-01; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Radiation Exposure; Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FPS 3-5 (Experimental): Frames per second are set at 3-5 at the beginning of the procedure
  Interventions: Radiation: frames per second
- FPS >5-8 (Experimental): Frames per second are set at >5-8 at the beginning of the procedure
  Interventions: Radiation: frames per second

INTERVENTIONS:
Radiation: frames per second — Other settings for frames per second

SUMMARY:
In the medical world more and more procedures are performed with the use of ionizing radiation (x-ray), both diagnostic and therapeutic. The main and most known risk is the development of malignancies as a result of the use of ionizing radiation.

Purpose of this study: To examine the patient radiation dose (PRD) if the frames per second (FPS) are set differently during the five most performed endourological procedures where fluoroscopy is used (insertion/replacement of ureteral stent, (mini-)percutaneous nephrolithotomy (PCNL/PNL), ureterorenoscopy (URS) and extracorporeal shock wave lithotripsy (ESWL/SWL)) and to propose an acceptable PRD for these procedures in a multicentric study.

ELIGIBILITY:
Inclusion Criteria:

* all patients who receive insertion/replacement of ureteral stent, URS (flexible or semirigid), (mini-)PCNL (including ECIRS) or ESWL under fluoroscopic with or without ultrasonic guidance
* Only cases performed or directly supervised by experts

Exclusion Criteria:

* Bilateral cases
* Diagnostic ureterorenoscopies
* Antegrade ureteroscopies
* Procedures for Upper Tract Urothelial Carcinoma (UTUC)
* Procedures on children (aged <18 years)
* Pregnant women
* Abnormal urinary anatomy (e.g. ureteral duplication, pelvic kidney, bladder derivation, horseshoe kidney)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-18 (Estimated); Study Completion 2024-12-18 (Estimated)

PRIMARY OUTCOMES:
Dose limit | 1 year
  Dose limit for the PRD during the insertion or replacement of a ureteral stent, URS, PCNL and ESWL

SECONDARY OUTCOMES:
Difference in PRD | 1 year
  Difference in the PRD during the insertion or replacement of a ureteral stent, URS, PCNL and ESWL when the FPS are set to 3 to 5 compared to >5 to 8
PRD different centres | 1 year
  PRD differ between the different participating urologists and centres
PRD difference complicated cases | 1 year
  PRD difference between normal and complicated cases

CONTACTS AND LOCATIONS:
Overall Officials: Vincent De Coninck, MD, Principal Investigator — Universiteit Antwerpen
Locations (2):
- Belgium (2):
  - AZ Klina, Brasschaat, Antwerp
  - UZA, Edegem, Antwerp

IPD SHARING:
Plan to Share IPD: No
All data will be stored in RedCAP and will only be accessible by the principal investigator

DOCUMENTS (1):
  • Informed Consent Form (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT06384105/ICF_000.pdf